CLINICAL TRIAL: NCT01781052
Title: DAILY: Observational Description of Compliance for the Daily Ventavis® Use Via the Insight Program in Class III Pulmonary Arterial Hypertension Patients
Brief Title: Observational Description of Compliance for the Daily Ventavis Use Via the Insight Program in Class III Pulmonary Arterial Hypertension Patients
Acronym: DAILY
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16133; VE1210FR (Other: Company internal); 2011/00416 (Other: Company internal)
Record Dates: First submitted 2013-01-22; First posted 2013-01-31 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-12

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Iloprost Compliance
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Iloprost

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Ventavis (Iloprost, BAYQ6256)

INTERVENTIONS:
Drug: Ventavis (Iloprost, BAYQ6256) — Initial dose: 2.5 µg per inhalation session; 6-9 inhalations/day. Dose can be increased to up to 5.0 µg per inhalation session.

SUMMARY:
This prospective, non-interventional, multi-center study documents observational data on subjects under routine treatment of Pulmonary Arterial Hypertension, functional class III with inhaled Iloprost administered with I-Neb AAD (Adaptive Aerosol Delivery) device. The observation period for each subject covers a one year treatment period with inhaled Ventavis. For each subject, the investigator or a delegate collects data as defined in the case report form at an initial visit, routine follow-up visit at 6 months and final visit at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥18 years
* Newly Treated with Ventavis or treated with Ventavis for less than 6 months, with I Neb AAD device for the application, as described in the SmPC (Summary of Product Characteristics), complemented by the Insight
* With Pulmonary Arterial Hypertension, Group I of the Dana point Pulmonary Hypertension Classification.
* WHO (World Health Organization) /NYHA (New York Heart Association) Functional class III
* Able and willing to give written informed consent for participation in the study

Exclusion Criteria:

Key contra indications:

* Hypersensitivity to the active substance or to any of the excipients.
* Conditions where the effects of Ventavis on platelets might increase the risk of haemorrhage (e.g. active peptic ulcers, trauma, intracranial haemorrhage).
* Severe coronary heart disease or unstable angina;
* Myocardial infarction within the last six months;
* Decompensated cardiac failure if not under close medical supervision;
* Severe arrhythmias;
* Cerebrovascular events (e.g. transient ischaemic attack, stroke) within the last 3 months.
* Pulmonary hypertension due to venous occlusive disease.
* Congenital or acquired valvular defects with clinically relevant myocardial function disorders not related to pulmonary hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 years and diagnosed with PAH (Pulmonary Arterial Hypertension), WHO/NYHA functional class III, Group I of the Dana point Pulmonary Hypertension Classification and newly Treated with Ventavis or treated with Ventavis for less than 6 months, with I-Neb AAD device for the application.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-09-11 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2017-01-16 (Actual)

PRIMARY OUTCOMES:
Compliance for each subject assessed by the mean daily number of inhalations of Ventavis. | Up to 12 months

SECONDARY OUTCOMES:
Compliance for each subject assessed by the mean daily number of inhalations of Ventavis | Up to 6 months
Total distance (meters) walked within 6 minutes assessed by the 6 Minutes Walking Distance Test | 6 and 12 months
Dyspnea Borg Category Ration 10 Scale values | 6 and 12 months
Quality of Life (EQ5D and LPH [Living with Pulmonary Hypertension] questionnaires) | 6 and 12 months
Investigator and patient satisfaction in the use of I-neb Insight tool assessed by a five level likert scale | Up to 12 months
Population characteristics | At baseline
  sociodemography, clinical aspects, risk factors

OTHER OUTCOMES:
Adverse events | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, France